CLINICAL TRIAL: NCT04577404
Title: A Phase 3, Multi-center, Open-label, Safety Extension Study of Oral Edaravone Administered Over 96 Weeks in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Safety Extension Study of Oral Edaravone Administered in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1186-A03; 2020-000376-38 (EudraCT Number); jRCT2041200084 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Edaravone

STUDY DESIGN:
Intervention Model Description: Single Arm Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MT-1186 (Experimental): Oral Edaravone administered once daily for 10 days out of 14, followed by a 14-day drug- free period
  Interventions: Drug: MT-1186

INTERVENTIONS:
Drug: MT-1186 — Treatment cycles with daily dosing for 10 days out of a 14-day period, followed by a 14 day drug free period up to 96 weeks of treatment or until the drug is commercially available in that country.
  Other Names: Oral Edaravone

SUMMARY:
This is a Phase 3, international, multicenter, open-label, long-term extension study. The primary objective of this study is to evaluate the long-term safety and tolerability of oral edaravone in subjects with Amyotrophic Lateral Sclerosis (ALS) for up to 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide signed and dated informed consent form (ICF) to participate in the study. Subjects must be able (in the judgment of the Investigator) to understand the nature of the study and all risks involved with participation in the study.
2. Subjects must be willing to cooperate and comply with all protocol restrictions and requirements.
3. Subjects who successfully completed Study MT-1186-A01.

Exclusion Criteria:

1. Subjects of childbearing potential unwilling to use a highly effective method of contraception from Visit 1 until 3 months after the last dose of study medication.
2. Subjects who have a significant risk of suicide. Subjects with any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without a specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the C-SSRS at Visit
3. Subjects who are not eligible to continue in the study, as judged by the Investigator.
4. Subjects who are unable to take their medications orally or through a PEG/RIG tube.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (44):
- United States (13):
  - St. Joseph's Hospital and Medical Center (SJHMC) - Barrow Neurological Institute (BNI) - The Gregory W. Fulton ALS and Neuromuscular Disease Center, Phoenix, Arizona
  - Neuromuscular Research Center, Phoenix, Arizona
  - Woodland Research Northwest, Rogers, Arkansas
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - UF Health Cancer Center, Gainesville, Florida
  - Emory University - School of Medicine, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Neurology Associates, P.C - Lincoln, Lincoln, Nebraska
  - Wake Forest University Baptist Medical Center (WFUBMC) - The J. Paul Sticht Center on Aging and Rehabilitation, Winston-Salem, North Carolina
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - Texas Neurology, PA, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Heritage Medical Research Clinic - University Of Calgary, Calgary, Alberta
  - University of Alberta - Walter C Mackenzie Health Sciences Centre (WCM), Edmonton, Alberta
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- France (4):
  - CHU-Nice - Hopital Pasteur 2, Nice, Cedex 1
  - Centre Hospitalier Esquirol, Limoges, Marcland
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux
  - Hopital Pierre Wertheimer - Hopital Neurologique, Paris
- Germany (2):
  - Deutsche Klinik fuer Diagnostik, Wiesbaden, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
- Italy (3):
  - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan, Lombardy
  - Universita degli Studi di Torino - Centro Regionale Esperto Per La Sclerosi Laterale Amiotrofica (CRESLA), Turin, Piedmont
  - Fondazione Serena Onlus - Azienda Ospedaliera Niguarda Ca Granda - Centro Clinico Nemo (Neuro Muscular Omnicentre), Milan
- Japan (19):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Murakami Karindoh Hospital, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - National Hospital Organization Hokkaido Medical Center, Sapporo, Hokkaido
  - National Hospital Organization Iou National Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Kumamoto Saishun Medical Center, Koshi-shi, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical And Dental Hospital, Niigata, Niigata
  - Kansai Electric Power Hospital Recruiting, Fukushima-ku, Osaka-shi, Osaka
  - National Hospital Organization Toneyama Medical Center, Toyonaka-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Neurological Hospital, Fuchū, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Genge A, Pattee GL, Sobue G, Aoki M, Yoshino H, Couratier P, Lunetta C, Petri S, Selness D, Todorovic V, Sasson N, Hirai M, Takahashi F, Salah A, Apple S, Wamil A, Kalin A, Jackson CE. Safety Extension Study of Edaravone Oral Suspension in Patients With Amyotrophic Lateral Sclerosis for up to an Additional 96 Weeks of Treatment. Muscle Nerve. 2025 Sep;72(3):450-454. doi: 10.1002/mus.28451. Epub 2025 Jun 9. PMID 40485494

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-1186: MT-1186 105mg (2 weeks On/Off)
Period: Overall Study
Arm/Group | MT-1186
Started | 124
Completed | 49
Not Completed | 75
Not completed — Adverse Event | 31
Not completed — Death | 1
Not completed — Lack of Efficacy | 3
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 21
Not completed — Switched to commercial oral Edaravon etc. | 12

BASELINE CHARACTERISTICS:
Arm/Group | MT-1186
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.1)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 84
  From 65 to 84 years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 118
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Events of Treatment Emergency Adverse Events (TEAEs), Adverse Drug Reactions (ADRs), Severe TEAEs, TESEAs, TEAEs Leading to Discontinuation, Any TEAEs Leading to Death
Description: AEs that occurred on or after the first dose in the MT-1186-A03 will be summarized, which implies AE that occurred during MT-1186-A01 will not be summarized.
  * Severe TEAEs: TEAEs which was classified as severe for the severity were analyzed. The severity of TEAEs was classified according to the following criteria: Mild (The event is transient and easily tolerated by the subject.), Moderate: The event causes discomfort and interferes with the subject's general condition.), and Severe (The event causes considerable interference with the subject's general condition and may be incapacitating.)
  * TESAEs, which is Serious TEAEs, is the TEAEs when the patients outcome is death, life-threatening, hospitalization, or disability or permanent damage.
Time Frame: up to 96 Weeks
Measure: Number; unit: events
Arm/Group | MT-1186
Number analyzed (Participants) | 124
events
  Number of TEAEs | 616
  Number of ADRs | 17
  Number of severe TEAEs | 60
  Number of TESAEs | 75
  Number of TEAEs leading to discontinuation | 35
  Number of TEAEs leading to death | 19

2. Primary Outcome: Number of Subjects of Treatment Emergency Adverse Events (TEAEs), Adverse Drug Reactions (ADRs), Severe TEAEs, TESAEs, TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: AEs that occurred on or after the first dose in the MT-1186-A03 will be summarized, which implies AE that occurred during MT-1186-A01 will not be summarized.
Time Frame: up to 96 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MT-1186
Number analyzed (Participants) | 124
Participants
  Number of TEAEs | 113
  Number of ADRs | 12
  Number of severe TEAEs | 44
  Number of TESEAs | 52
  Number of TEAEs leading to discontinuation | 28
  Number of TEAEs leading to death | 19

3. Other Pre Specified Outcome: Change From Baseline of ALS Functional Rating Scale-Revised (ALSFRS-R) at Week 96
Description: ALS Functional Rating Scale- Revised (ALSFRS-R). The ALSFRS-R is rating scale (ratings 0 = can't do, to 4 = normal ability) used to determine participants' assessment of their capability and independence in 12 functional activities.
Time Frame: Baseline to Week 96
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Number of Events of Death, Tracheostomy, or Permanent Assisted Mechanical Ventilation
Time Frame: up to 96 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 96 weeks
Arm/Group | MT-1186
All-Cause Mortality (participants affected / at risk) | 19/124
Serious Adverse Events (participants affected / at risk) | 52/124
Other Adverse Events (participants affected / at risk) | 70/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 (N=124)
Pneumonia (Infections and infestations) | 3
Pneumonia staphylococcal (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Assisted suicide (Psychiatric disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 6
Subarachnoid haemorrhage (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Myocarditis (Cardiac disorders) | 1
Phlebitis (Vascular disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 7
Ileus paralytic (Gastrointestinal disorders) | 1
Aerophagia (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Accidental death (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Gastrostomy (Surgical and medical procedures) | 2
Device malfunction (Product Issues) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 (N=124)
Constipation (Gastrointestinal disorders) | 16
Dysphagia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 7
COVID-19 (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 8
Fall (Injury, poisoning and procedural complications) | 20
Muscular weakness (Musculoskeletal and connective tissue disorders) | 18
Dysarthria (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT04577404/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT04577404/SAP_001.pdf